CLINICAL TRIAL: NCT06120205
Title: SELF-CERV Pivotal Study: Method Comparison of Self-collection Using the Teal Wand Self-Collection Device and HCP (Health Care Provider) Cervical Collection for Detection of High-risk HPV (hrHPV) for Cervical Cancer Screening
Brief Title: SELF-CERV Pivotal Study: SELF-Collection for CERVical Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teal Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CLN-TP-020
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Hpv; HPV 16 Infection; HPV Infection; High Risk HPV
Keywords: screening; self-collect; HPV; cervical cancer screening
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Self-Collection / Clinician Collection (Other): Patient serves as own comparator/control in this method comparison study where the investigational intervention is use of the self-collect device and the comparator is the standard of care clinician collection.
  Interventions: Device: Teal Wand Self-Collection Device Group

INTERVENTIONS:
Device: Teal Wand Self-Collection Device Group — Participants will use the Instructions for Use to perform self-collection of vaginal cells and material using the Teal Wand Self-Collection Device, and will fill out a usability survey and a satisfaction and needs survey. A healthcare provider collected sample will be performed by a clinician after self-collection. The patient will serve as their own comparator/control.
  Other Names: Clinician Collection

SUMMARY:
The goal of this method comparison study is to compare the detection of hrHPV collected using the Teal Wand Self-Collection device to hrHPV detected from HCP (health care provider) cervical collection using primary HPV testing assays.

Participants will be asked to use the Teal Wand to provide a self-collected sample prior to a healthcare provider collected sample to be tested for hrHPV. Secondary measure will include usability and preferences.

DETAILED DESCRIPTION:
To demonstrate that participants who are representative of the intended use population can understand the Instructions for Use (IFU) and appropriately use the Teal self-collection device to collect adequate vaginal cells/material for use in primary hrHPV screening (primary outcome).

To produce sufficient primary hrHPV test results following self-collection, as compared to the current SoC method of HCP specimen collection, when paired samples are tested using FDA approved primary hrHPV assays (Roche cobas and/or BD OnClarity).

Primary Effectiveness Objective

• To evaluate the performance of a self-collect device for hrHPV detection as compared to standard of care (SoC) by:

* Agreement of hrHPV self-collected sample(s) as compared to HCP-collected sample results.
* Calculating the invalid rate of tested samples.

ELIGIBILITY:
Group 1: Inclusion Criteria - General Population Group

1. Participant is 25 to 65 years of age and willing to provide informed consent.
2. Participant has an intact cervix.

Group 2: Inclusion Criteria - Enriched Population Group

1. Participant is 25 to 65 years of age and willing to provide informed consent.
2. Participant has an intact cervix.
3. One or more of the below:

   * Prior diagnosis of hrHPV within previous 6 months and/or
   * Positive cervical Pap cytology result (ASCUS, ASC-H, LSIL, HSIL, SCC, AIS) within previous 6 months and/or
   * Presenting for colposcopy/LEEP/excisional intervention

Exclusion Criteria - All Groups

1. Participant has impaired decision-making capacity or is unable to provide informed consent.
2. Participant has undergone partial or complete hysterectomy including removal of the cervix.
3. Participant on whom any form of cervical tissue alteration or surgery has been performed within the prior < 5 months, including: conization, loop electrosurgical excision procedure (LEEP), laser ablative surgery, or cryotherapy.
4. Participant is pregnant (based on self-reporting).
5. Participant who reports or is experiencing menstrual bleeding.
6. Participant is participating in another clinical study for an investigational device, drug, or biologic that, in the investigator's opinion, would interfere with the results of this study.
7. Any medical reason that, in the investigator's judgment, would disqualify the participant for a routine pelvic exam with cervical sample collection.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Detection of hrHPV in self-collect and clinician collect samples | Samples tested within 7 days of collection
  PPA/NPA (Positive Percent Agreement)/(Negative Percent Agreement) of hrHPV detection of self-collected and clinician collected samples
Safety: SAE rate | 6-14 days following collections
  SAE rate is equivalent for both self-collect and clinician collect interventions

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Birmingham OBGYN / Alabama Clinical Therapeutics, Birmingham, Alabama
  - Planned Parenthood Northern California, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Planned Parenthood Southern New England, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Woman's Hospital, Baton Rouge, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Planned Parenthood League of Massachusetts, Boston, Massachusetts
  - Planned Parenthood St. Louis Region, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - New York University Langone Hospital, Mineola, New York
  - Unified Women's Clinical Research Raleigh, Raleigh, North Carolina
  - Unified Women's Clinical Research - Lyndhurst, Winston-Salem, North Carolina
  - Planned Parenthood Gulf Coast, Houston, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
De-identified results only

REFERENCES:
- [Background] Onabolu AO, Oluwole OS, Bokanga M. Loss of residual cyanogens in a cassava food during short-term storage. Int J Food Sci Nutr. 2002 Jul;53(4):343-9. doi: 10.1080/09637480220138151. PMID 12090030
- [Derived] Fitzpatrick MB, Behrens CM, Hibler K, Parsons C, Kaplan C, Orso R, Parker L, Memmel L, Collins A, McNicholas C, Crane L, Hwang Y, Sutton E, Coleman J, Kuroki L, Harshberger K, Williams S, Jennings A, Buccini F, Gillis L, Novetsky AP, Hawkes D, Saville M, Depel T, Aviki E, Sheth SS, Conageski C. Clinical Validation of a Vaginal Cervical Cancer Screening Self-Collection Method for At-Home Use: A Nonrandomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e2511081. doi: 10.1001/jamanetworkopen.2025.11081. PMID 40388167